CLINICAL TRIAL: NCT06947525
Title: Effects of Shotblocker and Manual Pressure on Pain and Satisfaction During Peripheral Venous Catheter Placement: A Randomized Controlled Trial
Brief Title: Effects of Shotblocker and Manual Pressure on Pain and Satisfaction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Serpil SU, Lecturer, PhD, RN, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NecErUn
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Pain; Satisfaction
MeSH Terms: conditions — Pain; Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual pressure (Experimental): Before placing a peripheral intravenous catheter in the manual pressure group, the vein entry area will be pressed with the right thumb for 10 seconds. The pressure will be applied until the nail bed turns white.
  Interventions: Other: Manual pressure
- Shotblocker (Experimental): In the Shotblocker group, the shotblocker will be placed 2 cm above the vein entry point and will remain throughout the procedure.
  Interventions: Other: Shotblocker
- Control (No Intervention): The control group will undergo standard peripheral catheter placement without any intervention.

INTERVENTIONS:
Other: Manual pressure — Before the procedure in the manual pressure group, the vein entry area will be pressed with the right hand thumb for 10 seconds. The pressure will be applied until the nail bed turns white.
  Arms: Manual pressure
Other: Shotblocker — In the Shotblocker group, the shotblocker will be placed 2 cm above the vein entry point and will remain throughout the procedure.
  Arms: Shotblocker

SUMMARY:
This study aims to determine the effects of shotblocker and manual pressure applied during peripheral venous catheter placement on pain and satisfaction. 81 patients hospitalized in the Urology clinic will be included in the study. Patients will be assigned to three groups as shotblocker (n=27), manual pressure (n=27) and control group (n=27) by block randomization method.

Research Hypotheses

* H1-1: The mean pain scores of the intervention group to which shotblocker was applied during peripheral intravenous catheterization are different from the control group.
* H1-2: The mean pain scores of the intervention group to which manual pressure was applied during peripheral intravenous catheterization are different from the control group.
* H1-3: The mean satisfaction scores of the intervention group to which shotblocker was applied during peripheral intravenous catheterization are different from the control group.
* H1-4: The mean satisfaction scores of the intervention group to which manual pressure was applied during peripheral intravenous catheterization are different from the control group.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the urology clinic,
* No verbal, perceptual and visual communication problems,
* Between the ages of 18 and 65,
* Literate,
* Volunteer to participate in the study,
* Not using medication that will create a chronic analgesic effect,
* Not having chronic or acute pain,
* No intervention has been performed on the vein where the PIC is placed in the last month,
* No scar tissue or infection in the areas where the PIC will be placed,
* Not having a disease that will cause problems in feeling pain (such as neuropathy)

Exclusion Criteria:

* The individual wants to leave the study,
* Feels unwell during the PIC placement (such as dizziness, palpitations),
* Uses sedatives or alcohol,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | The peripheral venous catheter will be filled within 1 minute after insertion.
  The minimum score on the scale is 0 and the maximum score is 10. A score of 0 indicates no pain, while a score of 10 indicates unbearable pain.

SECONDARY OUTCOMES:
Patient Satisfaction Scale | The peripheral venous catheter will be filled within 1 minute after insertion.
  It is a horizontal scale that can be scored between 0 and 10. It is a measurement tool that starts with "I am not satisfied at all - 0" - "I am very satisfied - 10" and ends with.The minimum score on the scale is 0 and the maximum is 10. A score of 0 indicates that the procedure is not satisfactory at all, while a score of 10 indicates that the procedure is very satisfactory.

IPD SHARING:
Plan to Share IPD: No